CLINICAL TRIAL: NCT01847794
Title: Clinical Significance of HER2 Positive Circulating Tumor Cells(CTCs) in the Peripheral Blood of Patients With Advanced Gastric Cancer
Brief Title: HER2 Positive CTC in Advanced Gastric Cancer
Acronym: AGC-HER2CTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CGOG5002
Record Dates: First submitted 2013-04-29; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: HER2 Positive Advanced Gastric Cancer

ARMS (1):
- chemotheropy (Experimental)
  Interventions: Device: Cell Search® CTC epithelial kit

INTERVENTIONS:
Device: Cell Search® CTC epithelial kit — Collect peripheral blood sample of 50 gastric cancer patients pre-chemotherapy and post two cycles of chemotherapy(response evaluation).
  Blood samples will be transferred to central lab to detect HER2 positive CTCs by Cellsearch epithelial kit.
  Tumor response evaluation will be performed after two cycles of chemotherapy by CT/MRI based on RECIST. Clinical data, including tumor stage, metastastic organ, chemotherapy regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
To identify the correlation of HER2 expression in tissue and peripheral CTC. to identify the HER2 expression in CTCs with clinical prognosis in advanced/metastatic gastric cancer.

Confirm the presence of CTCs are sensitive for monitoring response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* HER2 overexpression confirmed by IHC or ISH (IHC 3+,or IHC2+/ISH+)
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥70
* Life expectancy of ≥3 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Previous systemic therapy for metastatic gastric cancer
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
HER2 positive CTC | 2 months

SECONDARY OUTCOMES:
clinical significance of HER 2 positive CTC | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD. PhD, Principal Investigator — Peking University
Locations (1):
- Peking cancer hospital, Beijing, Beijing Municipality, China